CLINICAL TRIAL: NCT06699342
Title: Pacing of Left Bundle Branch Area and Atroventricular Node ablatIon in Patients With Symptomatic Atrial Fibrillation
Acronym: PALLIATE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALLIATE-AF
Record Dates: First submitted 2024-11-03; First posted 2024-11-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; left bundle branch area pacing; Atrioventricular node ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LBBAP+AVNA arm (Experimental): Left bundle branch area pacing combined with atrioventricular node ablation.
  Interventions: Procedure: Pacemaker implantation with Left bundle branch area pacing (LBBAP); Procedure: Atrioventricular node ablation (AVNA)
- Control arm (Sham Comparator): Pharmacologic treatment optimized according to guidelines in patients with permanent atrial fibrillation refractory or intolerant to drug therapy or catheter ablation.
  Interventions: Drug: Pharmacologic therapy optimized for Atrial Fibrillation management

INTERVENTIONS:
Procedure: Pacemaker implantation with Left bundle branch area pacing (LBBAP) — Left bundle branch pacing is a novel pacing modality that can bypass the pathological or disease-vulnerable region in the cardiac conduction system, to provide physiological pacing modality for patients.
  The procedure involves the implantation of a permanent pacemaker with a pacing lead positioned at the left bundle branch area to achieve physiological conduction system pacing. LBBAP-Pacemaker device and leads should be implanted according to the physician's standard practice.
  Arms: LBBAP+AVNA arm
Procedure: Atrioventricular node ablation (AVNA) — Atrioventricular node ablation uses heat energy, called radiofrequency energy, to destroy the area between the upper and lower heart chambers. This area is called the atrioventricular node.
  Arms: LBBAP+AVNA arm
Drug: Pharmacologic therapy optimized for Atrial Fibrillation management — Pharmacologic therapy includes rate control with beta-blockers (e.g., bisoprolol), calcium channel blockers (e.g., diltiazem), or antiarrhythmic drugs (e.g., flecainide, propafenone, dronedarone, amiodarone) along with anticoagulation therapy (e.g., apixaban) as per current clinical guidelines (e.g., ESC 2024 or ACC/AHA/HRS 2023) in patients with permanent atrial fibrillation refractory or intolerant to drug therapy or catheter ablation.
  Treatment is tailored based on patient tolerance and clinical efficacy.
  Arms: Control arm

SUMMARY:
This study aimed to compare the clinical outcomes of left bundle branch area pacing combined with atrioventricular node ablation and pharmacologic treatment optimized according to guidelines in patients with symptomatic atrial fibrillation refractory or intolerant to drug therapy or catheter ablation.

DETAILED DESCRIPTION:
* Multicenter, randomized, open-label clinical trial
* Randomization 1:1 fashion A randomly permuted-block randomization list was generated by computer at a central location and was stratified by center.
* Study duration:

  1. 6 months (for primary outcome)
  2. 24 months (for secondary outcomes)
* Study subjects number: 50 patients (25 patients per group)
* Procedures

  * Atrioventricular node ablation after successful left bundle branch area pacing at the same procedure time.
  * Left bundle branch area pacing will be performed in all patients (using lumenless or stylet-driven lead, on the operator's discretion)
  * Atrioventricular node ablation will be performed using the quadripolar 7-Fr 3.5-mm tip ablation catheter and the use of 8.5-F sheath (SR0 or SL1, St. Jude Medical Inc., St. Paul, MN, USA) depending on the operator's experience, and if not stable or failed, a deflectable sheath (Agilis, Abbott Electrophysiology, Menlo Park, CA, USA) will be used. Repeated ablation procedures will be recommended during follow-up if regression of atrioventricular block has occurred.
  * Immediately after implant, devices were programmed to achieve the shortest QRS duration. Unipolar pacing was initially used to determine left bundle branch capture.

ELIGIBILITY:
Inclusion:

Patients who meet all of the following inclusion criteria 1)-6).

1. Permanent atrial fibrillation
2. Age ≥ 65 years
3. Refractory or intolerant to antiarrhythmic drugs, rate control medications, or catheter ablation
4. New York Heart Association (NYHA) functional class II- IV
5. LVEF > 40% (within the past 3 months)
6. Patients with at least one of the following:

   1. HF hospitalization (defined as HF as the major reason for hospitalization or treatment for HF lasting ≥12 hours and including treatment with intravenous (IV) diuretics at a healthcare facility) within 12 months
   2. Elevated NT-proBNP (>900 pg/ml) in the 30 days prior to enrollment

Exclusion:

Patients who meet at least one of the following exclusion criteria 1)-11).

1. Asymptomatic atrial fibrillation
2. Life expectancy to < 12 months.
3. Primary moderate to severe valvular disease (except for functional mitral valve regurgitation or tricuspid valve regurgitation)
4. Mechanical tricuspid valve replacement
5. Severe chronic kidney disease (estimated Glomerular Filtration Rate ≤ 15 ml/1,73 m2 or receiving renal replacement treatment including hemodialysis or peritoneal dialysis)
6. Obstructive hypertrophic cardiomyopathy
7. Infiltrative cardiomyopathy (amyloidosis, sarcoidosis, Fabry disease, others)
8. Acute coronary syndrome or coronary revascularization (CABG or PCI) <3 months
9. Severe primary pulmonary disease such as cor pulmonale, irreversible lung disease requiring inhalers, oxygen supplementation
10. Pacemaker/ICD/CRT treatment ongoing, or current pacemaker indication
11. Simultaneous participation in a different randomized clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP concentration (pg/ml) from baseline to 6-month follow-up | 6 months after intervention.

SECONDARY OUTCOMES:
Change in NT-proBNP concentration (pg/ml) at 12, and 24 months | 12 months and 24 months after intervention.
Change in health-related quality of life measured by 36-item short form survey (SF-36) questionnaire at 6, 12, 24 months | 6, 12 and 24 months after intervention.
  The SF-36 is a 36-item questionnaire that measures health-related quality of life across eight domains, including physical functioning, bodily pain, and mental health. Scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Change in health-related quality of life measured by EuroQol 5-Dimension Questionnaire (EQ-5D) at 6, 12, 24 months | 6, 12 and 24 months after intervention.
  The EuroQol 5-Dimension Questionnaire (EQ-5D) evaluates health-related quality of life using a descriptive system with five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores are derived as an index value (range: -0.594 to 1)
  The value attached to an EQ-5D profile according to a set of weights that reflect, on average, people's preferences about how good or bad the state is. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'
Change in left ventricular ejection fraction (LV-EF, %) at 6, 12, and 24 months | 6, 12 and 24 months after intervention
Change in left ventricular end-diastolic diameter (LVEDD, mm) at 6, 12, and 24 months | 6, 12 and 24 months after intervention.
Change in left ventricular end systolic diameter (LVESD, mm) at 6, 12, and 24 months | 6, 12 and 24 months after intervention.
Change in New York Heart Association (NYHA) functional class at 6, 12, and 24 months | 6, 12 and 24 months after intervention.
  The NYHA functional classification system assesses the severity of heart failure symptoms on a scale from Class I (best) to Class IV (worst). Changes in functional class will be evaluated at 6, 12, and 24 months after the intervention to determine the impact on patients' physical activity and symptom burden.
Change in 6 min walk test at 6, 12, and 24 months | 6, 12, and 24 months after intervention
Change in cognitive function measured by Montreal Cognitive Assessment (MoCA) score at 6, 12, and 24 months | 6, 12 and 24 months after intervention.
  The Montreal Cognitive Assessment (MoCA) is a widely used cognitive screening tool that assesses various cognitive domains, including memory, attention, language, visuospatial skills, and executive function. The MoCA score ranges from 0 to 30, with higher scores indicating better cognitive function. A score of 26 or above is generally considered normal, while lower scores suggest cognitive impairment. Changes in MoCA scores will be evaluated at 6, 12, and 24 months post-intervention.
Procedure-related complications (tamponade, device infection, re-intervention, pneumothorax, vascular complications, others) | 24 months after intervention.
The all-cause mortality at 24 months | 24 months after intervention.
  Death from any cause during the 24-month follow-up period.
Worsening Heart Failure (HF) at 24 Months | 24 months after intervention.
  *Worsening HF with or without hospitalization: symptoms, signs, imaging, and analytical criteria that require unplanned medical attention with an increase of diuretic use, intravenous diuretic therapy
Composite Outcome: Mortality and worsening heart failure (HF) at 24 months | 24 months after intervention.
  Participants meeting at least one of the criteria: (a) all-cause mortality, (b) worsening heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea